CLINICAL TRIAL: NCT03563443
Title: Evaluation of Genomic Imprinting Testing for Detection and Surveillance of Bladder Cancer Patients
Brief Title: Genomic Imprinting Testing for Diagnosis of Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: LiSen imprinting diagnostic (LSID) Company (Unknown)
Responsible Party: Principal Investigator, Zeng Shuxiong, M.D., Ph.D, Changhai Hospital
Other Study IDs: CH-urology-bladder marker-001
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Bladder Cancer; Urine Marking; Diagnoses Disease
Keywords: Bladder Cancer; Genomic imprinting; Urine biomarker; Diagnosis; Surveillance
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Loss of imprinting and Copy number variation (LOI & CNV) is epigenetic change that the silenced copy of an imprinting gene is activated through demethylation. Numerous studies indicate that LOI exists ubiquitously in cancers and precede morphological changes. In contrast, LOI rarely happens in normal somatic cells. Therefore, the methylation status of imprinting genes can act as a biomarker to detect and analyze the abnormal cast-off cells in urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder cancer patients: Diagnosed bladder cancer patients who are being monitored will be the experimental group to develop the LOI panel, and subsequent cohort will be used to confirm the sensitivity and specificity of this urinary analysis.
  Interventions: Diagnostic Test: Genomic Imprinting Testing
- Non-cancer participants: Patients being treated for other diseases but without any tumor or healthy participants will provide a negative control to provide data for developing the LOI diagnostic panel
  Interventions: Diagnostic Test: Genomic Imprinting Testing

INTERVENTIONS:
Diagnostic Test: Genomic Imprinting Testing — The changes of LOI The obtained LOI from morning urine and tumor will be tested by LiSen imprinting diagnostic (LSID)

SUMMARY:
Urine analysis provide a promising non-invasive liquid biopsy for diagnosis of bladder cancer. Molecular biomarkers in urine may serve as important diagnostic and prognostic indicators for bladder cancer. Many alterations of genes and proteins have been identified in the urinary for diagnosis of bladder cancer. However, not all bladder cancer patients have the same alterations due to tumor heterogeneity. Thus, to reach satisfactory sensitivity and specificity a new diagnostic molecular alteration should exists ubiquitously in cancers. Numerous studies indicate that Loss of imprinting (LOI) exists ubiquitously in cancers and precede morphological changes. The investigators will conduct a prospective evaluation of a panel of LOI changes in urine test for detection and surveillance of bladder cancer patients.

DETAILED DESCRIPTION:
During the progression of tumor, molecular changes in both genomics and epigenomics occur prior to morphological changes in cells and tissues, therefore molecular biological test is more sensitive to detect cancer at early stage. Genomic imprinting is one kind of epigenetic regulation that controls gene expression. In detail, a copy of gene on the certain maternal or paternal allele is silenced through methylation, while the other acts normally. This kind of genes are named imprinting genes. Loss of imprinting and Copy number variation (LOI & CNV) is epigenetic change that the silenced copy of an imprinting gene is activated through demethylation. Numerous studies indicate that LOI exists ubiquitously in cancers and precede morphological changes. In contrast, LOI rarely happens in normal somatic cells. Therefore, the methylation status of imprinting genes can act as a biomarker to detect and analyze the abnormal cells.

The investigators will develop a couple of common LOI to establish a predictive diagnostic LOI panel in urine with optimal and robust efficacy in diagnosis of bladder cancer by analyzing LOI in urine from bladder cancer patients and control group that without any tumor in urinary system or other organs. Moreover, the changes of LOI in urine collected before and 1 year after transurethral resection of non-muscle invasive bladder cancer (NIMBC) will also be monitored. External consistency validation will be performed on subsequent urine from patients and control participants collection.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients diagnosed with of bladder cancer by cystoscopy and biopsy. 2. Participants without any tumor disease and willing to attend the study by providing morning urine.

3. Moring urine and available tumor tissue obtained by biopsy. 4. Male or female patients aged >= 18 years. 5. Participants signed informed consent form.

Exclusion Criteria:

- 1. Age under 18 years 2. Individuals unwilling to sign the IRB-approved consent form and unwilling to follow the protocol to submit the serial urine for test after surgery 3. Comorbidities that will prohibit or make serial urine collection and cystoscopic examination difficult or impossible during follow up.

4. Prior diagnosis of cancer except bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer or participants in control group in Changhai Hospital from December 2017 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of urinalysis by LOI urine analysis | In the middle of the study, an average of 12 months
  Number of patients "declared positive" with the LOI urine test among the patients suffered from bladder cancer
Specificity of urinalysis by LOI urine analysis | In the middle of the study, an average of 12 months
  Number of patients "declared negative" with the LOI urine test among the patients who are without cancer

SECONDARY OUTCOMES:
Identification of sensitivity of urinalysis by LOI urine analysis to predict the recurrence of bladder cancer within 1 year after transurethral resection of NMIBC | Through study completion, an average of 24 months
  Number of patients "declared positive" with the LOI urine test after bladder cancer surgery among the patients being confirmed to have bladder cancer by cystoscopic examination and biopsy
Identification of specificity of urinalysis by LOI urine analysis to predict the free of bladder cancer recurrence within 1 year after transurethral resection of NMIBC | Through study completion, an average of 24 months
  Number of patients "declared negative" with the LOI urine test after bladder cancer surgery among the patients being confirmed to have no bladder cancer recurrence by cystoscopic examination
Comparison of the sensitivity of the urine LOI analysis versus urine cytology | In the middle of the study, an average of 12 months
  Number of patients "declared positive" with the LOI analysis versus patients "declared positive" with the urine cytology
Comparison of the specificity of the urine LOI analysis versus urine cytology | In the middle of the study, an average of 12 months
  Number of patients "declared negative" with the LOI analysis versus patients " declared negative " with the urine cytology

CONTACTS AND LOCATIONS:
Overall Officials: Chuangliang Xu, M.D., Ph.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelinic P, Shaw P. Loss of imprinting and cancer. J Pathol. 2007 Feb;211(3):261-8. doi: 10.1002/path.2116. PMID 17177177
- [Background] Haig D. Maternal-fetal conflict, genomic imprinting and mammalian vulnerabilities to cancer. Philos Trans R Soc Lond B Biol Sci. 2015 Jul 19;370(1673):20140178. doi: 10.1098/rstb.2014.0178. PMID 26056362
- [Background] Uribe-Lewis S, Woodfine K, Stojic L, Murrell A. Molecular mechanisms of genomic imprinting and clinical implications for cancer. Expert Rev Mol Med. 2011 Jan 25;13:e2. doi: 10.1017/S1462399410001717. PMID 21262060
- [Background] Jirtle RL. Genomic imprinting and cancer. Exp Cell Res. 1999 Apr 10;248(1):18-24. doi: 10.1006/excr.1999.4453. PMID 10094809